CLINICAL TRIAL: NCT04952441
Title: A Randomized Controlled Trial of the RISE Program for Nurses
Brief Title: RISE Program for Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1361876
Record Dates: First submitted 2021-06-17; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into either the intervention group or the wait-list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group will attend the RISE program which consists of eight 90-minute weekly psychoeducational group sessions facilitated by a licensed mental health counselor
  Interventions: Behavioral: RISE Program
- Wait-list Control Group (Active Comparator): The control group will attend the RISE program after the 3 month wait-list period (study months 6-7)
  Interventions: Behavioral: RISE Program

INTERVENTIONS:
Behavioral: RISE Program — Psychoeducational sessions designed to impact Resilience, Insight, Self-Compassion, and Empowerment

SUMMARY:
The purpose of this study is to determine whether the RISE program has a significant impact on nurses' resilience, insight, self-compassion, and empowerment, as well as mental and physical well-being, in their personal lives and their working environment.

DETAILED DESCRIPTION:
This study will include the face-to-face visits of eight weekly 90-minute psychoeducational group sessions in a private conference room at AdventHealth. No absences are permitted due to lack of engagement. Participants will only be compensated for the number of attended sessions. The LMHC facilitator will send a reminder email to the control group participants after the intervention group participants attend their eighth session.

There will be three unpaid optional follow-up monthly booster sessions that focus on skill development. Participants will be invited to attend these booster sessions during the 3 months following their group's RISE Program. Attendance will be recorded. No other data will be collected during the booster sessions.

The following assessments will be used to measure study outcomes: Brief Resilience Scale (BRS); Self-Reflection and Insight Scale (SRIS); Self-Compassion Scale - Short Form (SCS-SF); Psychological Empowerment Instrument (PEI); Stress Mindset Measure - General (SMM-G); Perceived Stress Survey (PSS); Maslach Burnout Inventory (MBI); Public Health Surveillance - Wellbeing Scale (PHS-WB); RAND MOS Sleep Scale Survey; RAND 36-Item Short Form Health Survey (SF-36); World Health Organization Health and Work Performance questionnaire (WHO-HPQ); and Work Productivity and Activity Impairment (WPAI) questionnaire. In addition, demographic assessments will be collected. Employment with AdventHealth will also be tracked longitudinally at 12 months with Human Resources.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years old
2. Licensed as an RN
3. RN employed by AdventHealth in a hospital-based setting at the Altamonte, Apopka, Celebration, Daytona Beach, DeLand, East, Fish Memorial, Kissimmee, New Smyrna Beach, Orlando, Palm Coast, Waterman, or Winter Park campus
4. Able to speak, read, and understand English fluently
5. Able to provide informed consent
6. Willing and able to comply with all study procedures and requirements for the duration of the study.

Exclusion Criteria:

1. Employed as an ARNP
2. Employed in a role that completes another RN's annual evaluations
3. A participant of the study in IRBNet #1234568 or IRBNet #1256670
4. At imminent risk of harm to themselves or others.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Self-Reflection and Insight Scale (SRIS) | Change from Baseline to 3 month follow up
  Participants will respond to a 20-item questionnaire using a 6-point scale where 1=Strongly disagree and 6=Strongly agree.

SECONDARY OUTCOMES:
Measure Name: Brief Resilience Scale (BRS) | Change from Baseline to 3 month follow up
  Participants will respond to a 6-item questionnaire measuring resilience. Responses will be provided on the following 5-point scale: 1=Strongly Disagree, 2=Disagree, 3=Neutral, 4=Agree, 5=Strongly Agree.
Self-Compassion Scale - Short Form (SCS-SF) | Change from Baseline to 3 month follow up
  Participants will respond to a 12-item questionnaire, indicating how often certain behaviors are personally experienced when in difficult times. Responses are provided on 5-point scale in which 1=Almost never and 5=Almost always.
Psychological Empowerment Instrument (PEI) | Change from Baseline to 3 month follow up
  Participants will respond to a 12-item questionnaire to items regarding self-orientations people may have with regard to their work role. Responses are provided on the following 7-point scale: 1=Very strongly disagree, 2=Strongly disagree, 3=Disagree, 4=Neutral, 5=Agree, 6=Strongly Agree, 7=Very Strongly Agree.
Stress Mindset Measure - General (SMM-G) | Change from Baseline to 3 month follow up
  Participants will respond to an 8-item questionnaire measuring stress. Responses will be provided on the following 5-point scale: 0=Strongly Disagree, 1=Disagree, 2=Neither Agree nor Disagree, 3=Agree, 4=Strongly Agree.
Perceived Stress Scale (PSS) | Change from Baseline to 3 month follow up
  Participants will respond to a 10-item questionnaire measuring perceived stress. Responses will be provided on the following 5-point scale: 0=Never, 1=Almost Never, 2=Sometimes, 3=Fairly Often, 4=Very Often.
Maslach Burnout Inventory Human Services Survey (MBI-HSS) for Medical Personnel (MP) | Change from Baseline to 3 month follow up
  Participants will respond to a 22-item questionnaire measuring burnout. Responses will be provided on the following 7-point scale: 0=Never, 1=A few times a year or less, 2=Once a month or less, 3=A few times a month, 4=Once a week, 5=A few times a week, 6=Everyday.
Public Health Surveillance - Wellbeing Scale (PHS-WB) | Change from Baseline to 3 month follow up
  Participants will respond to a 10-item questionnaire measuring perception of personal well-being and satisfaction. Responses will be provided on a 5-point scale (6 items) and a 10-point scale (4 items).
RAND Medical Outcomes Study (MOS) Sleep Scale Survey | Change from Baseline to 3 month follow up
  Participants will respond to a 12-item questionnaire with self-reported information related to sleep patterns. Responses will be provided on the following 6-point scale: 1=All of the time, 2=Most of the time, 3=A good bit of the time, 4=Some of the time, 5=A little of the time, 6=None of the time.
RAND 36-Item Short Form Health Survey (SF-36) | Change from Baseline to 3 month follow up
  Participants will respond to a 36-item questionnaire with self-reported health ratings and perceived impact of one's health on a variety of daily activities. Response options for questionnaire items vary from 3-point scale, 5-point scale, and Yes/No responses.
Absenteeism and Presenteeism questions of the World Health Organization's Health and Work Performance Questionnaire (WHO-HPQ) | Change from Baseline to 3 month follow up
  Participants will respond to 11 absenteeism and presenteeism questions abstracted from the full HPQ. Responses for 2 items require self-reported information regarding hours worked and hours the employer expects the participant to work in 7 days. 6 items require participants to provide work experience information from the past 4 weeks. Responses for 3 items are provided on a 10-point scale in which 0=Worst Performance, and 10=Top Performance. Responses are input into a provided formula for scoring; a higher absenteeism score indicates higher amount of absenteeism, while a higher presenteeism score indicates lower amount of lost performance.
Work Productivity and Activity Impairment Questionnaire (WPAI) | Change from Baseline to 3 month follow up
  Participants will respond to a 6-item questionnaire, answering questions about the perceived effect of personal health problems on one's ability to work or perform activities. Responses are provided in a Yes/No format or using a 10-point scale in which 0=Health problems had no effect on my work and 10=Health problems completely prevented me from working.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Sawyer, PhD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth, Orlando, Florida, United States

REFERENCES:
- [Background] Acker KH. Do critical care nurses face burnout, PTSD, or is it something else?: getting help for the helpers. AACN Clin Issues Crit Care Nurs. 1993 Aug;4(3):558-65. PMID 8136229
- [Background] Bann CM, Kobau R, Lewis MA, Zack MM, Luncheon C, Thompson WW. Development and psychometric evaluation of the public health surveillance well-being scale. Qual Life Res. 2012 Aug;21(6):1031-43. doi: 10.1007/s11136-011-0002-9. Epub 2011 Sep 23. PMID 21947657
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Crum AJ, Salovey P, Achor S. Rethinking stress: the role of mindsets in determining the stress response. J Pers Soc Psychol. 2013 Apr;104(4):716-33. doi: 10.1037/a0031201. Epub 2013 Feb 25. PMID 23437923
- [Background] Kessler RC, Barber C, Beck A, Berglund P, Cleary PD, McKenas D, Pronk N, Simon G, Stang P, Ustun TB, Wang P. The World Health Organization Health and Work Performance Questionnaire (HPQ). J Occup Environ Med. 2003 Feb;45(2):156-74. doi: 10.1097/01.jom.0000052967.43131.51. PMID 12625231
- [Background] Mealer ML, Shelton A, Berg B, Rothbaum B, Moss M. Increased prevalence of post-traumatic stress disorder symptoms in critical care nurses. Am J Respir Crit Care Med. 2007 Apr 1;175(7):693-7. doi: 10.1164/rccm.200606-735OC. Epub 2006 Dec 21. PMID 17185650
- [Background] Mealer M, Burnham EL, Goode CJ, Rothbaum B, Moss M. The prevalence and impact of post traumatic stress disorder and burnout syndrome in nurses. Depress Anxiety. 2009;26(12):1118-26. doi: 10.1002/da.20631. PMID 19918928
- [Background] Mealer M, Conrad D, Evans J, Jooste K, Solyntjes J, Rothbaum B, Moss M. Feasibility and acceptability of a resilience training program for intensive care unit nurses. Am J Crit Care. 2014 Nov;23(6):e97-105. doi: 10.4037/ajcc2014747. PMID 25362680
- [Background] Mealer M, Jones J, Newman J, McFann KK, Rothbaum B, Moss M. The presence of resilience is associated with a healthier psychological profile in intensive care unit (ICU) nurses: results of a national survey. Int J Nurs Stud. 2012 Mar;49(3):292-9. doi: 10.1016/j.ijnurstu.2011.09.015. Epub 2011 Oct 5. PMID 21974793
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Hughes RG, editor. Patient Safety and Quality: An Evidence-Based Handbook for Nurses. Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK2651/ PMID 21328752
- [Background] Grant AM, Franklin J, Langford P. The Self-Reflection and Insight Scale: A new measure of private self-consciousness. Social Behavior and Personality. 2002; 30(8): 821-836
- [Background] Maslach C, Jackson SE, Leiter MP. (1996). Maslach Burnout Inventory manual (3rd ed.). Palo Alto, CA: Consulting Psychologists Press
- [Background] Spreitzer GM. Psychological empowerment in the workplace: Dimensions, measurement, and validation. Academy of Management Journal. 1995; 38(5): 1442-1465